CLINICAL TRIAL: NCT06949345
Title: Health Literacy in Relation to Attitudes Towards Traditional and Complementary Medicine Among Physical Therapy and Rehabilitation Patients.
Brief Title: Health & Digital Literacy and Complementary Medicine Attitudes in Rehabilitation Patients
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, PT, PhD, Karabuk University
Other Study IDs: health literacy and CAM
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-04

CONDITIONS: Health Literacy Level; Digital Health Literacy; Complementary and Alternative Therapies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of a Physical Medicine and Rehabilitation Clinic

SUMMARY:
This observational study aims to evaluate the relationship between health and digital health literacy and attitudes toward complementary and alternative medicine (CAM) in patients visiting a physical medicine and rehabilitation outpatient clinic. Low health literacy may lead patients to try potentially unsafe herbal products influenced by commercial or social media sources. This study highlights the importance of understanding patients' attitudes toward such methods and aims to contribute to the development of educational efforts to improve health literacy. Increasing patients' awareness can support better decision-making, enhance rehabilitation outcomes, and promote the use of evidence-based practices in physical medicine clinics..

DETAILED DESCRIPTION:
This observational, cross-sectional clinical study will be conducted in the Physical Medicine and Rehabilitation outpatient clinic of Karabük Training and Research Hospital. The target population includes at least 200 volunteer patients aged between 18 and 65 years. The primary objective is to evaluate the level of general and digital health literacy and the attitudes toward complementary and alternative medicine (CAM), and to investigate the relationship between these variables.

Participants will be recruited consecutively from the outpatient clinic. Inclusion criteria consist of being aged 18-65, literate, and volunteering to participate. Individuals who are unwilling or unable to cooperate, or who have cognitive or psychiatric impairments that may hinder questionnaire completion, will be excluded from the study.

Data will be collected through self-administered or interviewer-assisted questionnaires. The tools to be used are:

A structured sociodemographic data form (age, gender, education level, marital status, etc.),

Health Literacy Index (25 items), assessing general health literacy,

Digital Health Literacy Instrument (DHLI) (18 items, 6 subscales), evaluating digital health-related skills,

Complementary and Alternative Medicine Attitude Scale (CAMAS) (27 items, 3 subscales), measuring participants' attitudes toward CAM.

Data will be analyzed using IBM SPSS software. Normality of data distribution will be assessed with the Kolmogorov-Smirnov test. Depending on data characteristics, appropriate statistical tests such as Pearson or Spearman correlation, independent sample t-tests, and ANOVA will be applied. The study will also compare health and digital health literacy levels and CAM attitudes across different sociodemographic and clinical variables.

Findings from this study are expected to highlight gaps in patient knowledge and perceptions regarding CAM and digital health, potentially informing future educational strategies and supporting evidence-based clinical decision-making in rehabilitation settings.

ELIGIBILITY:
Inclusion Criteria:

* being aged 18-65
* being literate
* Volunteering to participate

Exclusion Criteria:

* Patients who are unwilling or unable to cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 65 years who are literate and voluntarily applying to the Physical Medicine and Rehabilitation outpatient clinic of Karabük Training and Research Hospital. Participants must be able to provide informed consent and complete the required questionnaires.
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Complementary, Alternative, Conventional Medicine Attitude Scale (CACMAS) | Baseline
  The CACMAS is a 27-item scale with three subscales: attitudes toward complementary, alternative, and conventional medicine.The scale uses a 7-point Likert-type rating system, with responses ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
  Total Score Range: 27 to 189 Interpretation: Higher scores indicate a more positive attitude toward the use of CAM and conventional medical practices.
Digital Health Literacy Instrument | Baseline
  The scale consists of 18 items across 6 dimensions: Information Seeking, Evaluation of Reliability, Determining Interest Level, Content Addition, Navigation Skills, and Privacy Protection. Participants rated their experiences on a 4-point Likert scale (1 = Very difficult, 2 = Difficult, 3 = Easy, 4 = Very easy) for the subdimensions of Information Seeking, Evaluation of Reliability, Determining Interest Level, and Content Addition. For Navigation Skills and Privacy Protection, a reverse-coded 4-point Likert scale was used (1 = Never, 2 = Occasionally, 3 = Rarely, 4 = Frequently). The overall and subscale scores ranged from 1 to 4, with scores below 2 indicating low digital health literacy, scores between 2 and 3 indicating moderate digital health literacy, and scores above 3 indicating high digital health literacy.
Health Literacy Scale | Baseline
  The HLS-25 is a 25-item instrument adapted into Turkish by Aras and Temel (2017) based on the simplified version of the Health Literacy Survey in Europe (HLS-EU). It consists of four subscales: accessing information (5 items, score range: 5-25), understanding information (7 items, range: 7-35), appraising information (8 items, range: 8-40), and applying information (5 items, range: 5-25).
  Total Score Range: 25 to 125 Interpretation: Higher scores indicate better health literacy. All items are scored on a 5-point Likert scale (1 = cannot do at all to 5 = no difficulty). There are no reverse-coded items. Lower scores reflect inadequate or problematic health literacy.

SECONDARY OUTCOMES:
Personal information form | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Metehan Yana, Study Chair — Karabuk University
Locations (1):
- Karabuk Education and Research Hospital, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Unal Toprak F, Coskun Palaz S, Caglar S. The impact of health literacy levels on women's fear of contracting Covid-19 and their attitudes toward holistic complementary and alternative medicine: Mediation analysis results. Health Care Women Int. 2023 Jul-Sep;44(7-8):869-884. doi: 10.1080/07399332.2022.2070623. Epub 2022 May 26. PMID 35616392
- [Background] Okawa Y, Ideguchi N, Yamashita H. Relationship between health literacy and attitudes toward acupuncture: A web-based cross-sectional survey with a panel of Japanese residents. PLoS One. 2023 Oct 20;18(10):e0292729. doi: 10.1371/journal.pone.0292729. eCollection 2023. PMID 37862311